CLINICAL TRIAL: NCT04339647
Title: Effect of the Community-based SIMS Programme on Preschool Children's Oral Hygiene Level: A Cluster Randomised Control Trial
Brief Title: Effect of the SIMS Programme on Preschool Children's Oral Hygiene Level
Acronym: SIMSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIRG035A
Record Dates: First submitted 2020-04-05; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Dental Plaque
Keywords: Preschool; Children; Dental plaque; Oral health behaviour; Health literacy
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Cluster Randomised Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The SIMS Programme (Experimental): The SIMS programme is a community-based intervention which improvised the usual care (defined as the existing preschool oral health programme) offered by the Ministry of Health. The target group is 5-6-year-old preschool children and their parents. Apart from the usual care, the 5-6-year-old children receive interventions carried out by teacher in school and home tooth brushing supervision by parents. In addition, parents/guardians will receive OHE from the DT team, free toothbrush and toothpaste (1000ppm F) for child home tooth brushing and supervised child home tooth brushing for 6 months.
  Interventions: Behavioral: The SIMS programme
- Control (No Intervention): The control group receives the usual care from the preschool oral health programme. The usual care is described as a DT team visiting the school to do an oral examination, provides OHE to the children, and applies fluoride varnish (20,000 ppmF) twice/year.

INTERVENTIONS:
Behavioral: The SIMS programme — The intervention targets 5-6-year-old preschool children and their parents. Apart from the usual care, 5-6-year-old children receive oral health lessons and supervised daily tooth brushing (1000ppm F) at school over a period of 6 months, as well as home tooth brushing supervision by parents for 6 months. Parents/guardians attend a meeting with a DT team at school to discuss on child's oral health status, receive OHE and free toothbrush and fluoride toothpaste (1000ppm F) for child home tooth brushing, and receive 10 oral health infographic messages from DT over a period of 5 months (with printed versions available).
  Arms: The SIMS Programme

SUMMARY:
This is a cluster randomised control trial targeting 5-6-year-old children and their parents in Kampar district, Perak, Malaysia for a period of 6 months. In total, 28 preschools are randomly assigned into intervention and control group (14 preschools per group). Sample size for each group is 317 children. The intervention group receives the SIMS programme (SIMSP) which is an improved version of the usual care, while the control group receives the usual care. Usual care in defined as the existing preschool oral health programme (POHP) offered by the Ministry of Health. The SIMSP is formulated based on the recommendations from the National Oral Health Survey of Preschool Children's (2015) report. It comprises active participation of dental therapists (DT), parents and class teachers in children's oral health. The concept of the SIMSP is that improvement in oral health behaviours and oral hygiene of preschool children would result in improvement of gingival health and caries level in their permanent teeth in the long term. On the other hand, the control group involves DT visiting preschools twice a year without parental nor teachers active involvement. The scientific hypothesis of the study is that the SIMSP is more effective to improve oral hygiene level of preschool children than the POHP over 6 months. The primary objective of the study is to assess the effect of the SIMSP versus the POHP in improving oral hygiene level among 5-6-year-old children over 6 months. The secondary objectives are to assess the changes in oral health behaviours among the children and oral health literacy among parents over 6 months.

DETAILED DESCRIPTION:
Study Design:

This is a cluster randomised controlled trial. The overall duration of the study is 9 months and the duration of the intervention is 6 months. The reporting of this study is done in accordance with the SPIRIT 2013 guidance for protocols of clinical trials and the CONSORT checklist.

Study setting:

The study involves government-funded preschools that receive the POHP in Kampar district, Perak, Malaysia. Based on this criteria, 53 preschools in Kampar district are eligible to be included in the study.

Randomisation:

The 53 preschools are paired according to geographical location and preschool characteristics into 24 pairs (5 preschools are not paired). Of the 24 pairs, 14 pairs are randomly selected using computer generated table. Subsequently, 2 preschools in each pair is randomly assigned to intervention and control group each using computer generated table.

Sample recruitment:

The study sample consists of 5-6-year-old preschool children from the 24 preschools and their parents. A written informed consent is obtained from parents and verbal agreement is obtained from children prior to the start of the study.

Sample size calculation:

Sample size calculation is based on the potential effect of the SIMSP to exert a small effect size dz = 0.30, α = 0.05, power = 0.8 on children's plaque score (primary outcome measure) and parental oral health literacy (OHL - secondary outcome measure) than the POHP over 6 months. Using G*Power version 3.1.9.2 software, the total number of sample is n = 352 (176 per group). Sample size calculation is also done based on the effect of the SIMSP to produce a 10% improvement (α = 0.05, power = 0.8) in child's oral health behaviours (OHB) than the POHP after 6 months. Using Power and Sample Size Calculation version 3.1.2 software, the total number of sample was n = 348 (174 per group). The highest total sample size (n = 352) is increased by 20% to account for non-respondents and multiplied by a design effect of 1.5 to produce final sample size, n = [352 + (352*0.2)] x 1.5 = 634 (317 per group).

Intervention:

The SIMSP, which refers to 'Program Senyuman Indah Milik Semua' in Malay, or 'The Beautiful Smile for All Programme' in English, consists of 3 components conducted by a dedicated team of DT (4 persons), parents, and preschool teachers. The target groups are preschool children and their parents/guardians. The content of the SIMSP is as follows:

Preschool children:

1. Oral examination by DT, oral health education (OHE) and fluoride varnish application twice/year (usual care/POHP);
2. In-school daily toothbrushing with fluoride toothpaste (1000ppm) supervised by the class teacher for 6 months;
3. Oral health lessons in class (including colouring worksheets) by the class teacher based on the Oral Health Education (OHE) booklet over a period of 6 months;
4. Home tooth brushing supervision by parents/guardians bedtime.

Parents/guardians:

1. Attend a meeting with DT at school to discuss on child's Caries Risk Assessment (CRA);
2. Receive OHE and diet counselling from DT based on child's CRA levels;
3. Receive free toothbrush and fluoride toothpaste (1000ppm) for child home tooth brushing;
4. Receive 10 oral health infographic messages from DT, delivered via electronic messaging application (WhatsApp) every 2 weeks for a duration of 5 months (printed leaflets delivered through class teacher for parents without a smartphone).

Control:

Oral examination by DT, oral health education (OHE), and fluoride varnish application twice/year (usual care/POHP).

Conduct of the study:

(A) Prior to intervention - development of the Oral Health Education booklet for teacher, training of teachers on its use, and development of oral health infographics for parents.

(B) Delivery of the intervention - the intervention is delivered in 3 phases;

Phase 1:

It involves an oral examination (including plaque assessment) of children in both groups by DT. On the same visit, a self-administered questionnaire is sent to parents through class teacher and collected after 1 week. Data in Phase 1 are baseline data for the study.

Phase 2:

This phase takes place 2 weeks after Phase 1. In the SIMSP, DT deliver OHE to children and apply fluoride varnish (20,000 ppmF) on their teeth. DT meet up with parents to discuss on child's CRA and provide OHE and diet counselling to parents according to their child's caries risk levels (low/medium/high). A set of free toothbrush and fluoride toothpaste (1000ppm fluoride) is distributed to parents for child's home use along with instructions on toothbrushing. Parents also receive 10 oral health infographics sent by DT via WhatsApp every 2 weeks for the next 5 months. Teachers are provided with the OHE booklet which contains 11 topics (and worksheets) to be used as a teaching aid to teach oral health lessons in class. Teachers are required to deliver 1 topic lesson every 2 weeks until all the 11 topics are delivered over 6 months. Teachers are also given enough supplies of toothbrush and fluoride toothpaste for children's tooth brushing after morning break at school over 6 months. Teachers are given a tooth model and instructions on toothbrushing by DT. In the control group, DT deliver OHE to children and apply fluoride varnish (20,000 ppmF) on their teeth.

Phase 3:

This phase takes place 24 weeks after Phase 2. In this phase, DT carry out restorative treatment on children using glass inomer cements followed by second application of fluoride varnish. This is carried out in both groups. The 6-month follow up for oral examination on children and parental questionnaire are carried out within 2 weeks after completion of Phase 3.

Monitoring the intervention:

The intervention is monitored by means of an activity book to be completed by DT, parents, and teachers, respectively throughout the 6 months. DT will tick off all activities that have been carried out at preschool in the 3 phases over the duration of 6 months. Accordingly, teachers will tick off the scheduled class lessons and daily toothbrushing activities. Parents will tick off the daily toothbrushing supervision of their children before bedtime. The activity books are reviewed periodically to assess for compliance. In terms of oral examination and parental questionnaire, those who are lost to follow up will not be replaced. Analysis will be by intention to treat.

Study tools:

1. A self-administered questionnaire consisting of 3 sections; (a) Demographics of the child and parents/guardians, (b) Child's oral health behaviours, and (C) The Malay version of Dental Health Literacy Assessment Instrument (Malay-DHLAI).
2. The Oral Cleanliness Index to assess plaque level.
3. The International Caries Detection and Assessment System (ICDAS) to assess caries.

Blinding:

This study uses a single-blinding strategy where the examiners who examine the children at baseline and 6-month follow up are blinded to the intervention group.

Calibration of examiners:

3 dental officers undergo calibration and standardisation on the use of ICDAS and Oral Cleanliness Index with a paediatric dentist. Calibration and standardisation are carried out at the Faculty of Dentistry, University of Malaya and again in field condition at one of the preschools not involved in the study. Inter- and intra-examiner reliability are assessed for both ICDAS and plaque score charting. Kappa score is used to assess agreement between and within examiners. For ICDAS, the inter-examiner Kappa scores ranged from 0.72-0.80 and the intra-examiner scores ranged from 0.70-0.84. For plaque scores, the inter-examiner Kappa scores ranged from 0.72-.80 and the intra-examiner scores ranged from 0.77-0.94.

Data management:

Data are checked after completion of oral examinations and after receiving the questionnaires. For any missing data, the child will be re-examined or the parents will be contacted again. Raw data are entered into Statistical Package for Social Science (SPSS) version 24.

Qualitative data collection:

Focus group discussions (FGD) with DT and preschool teachers are conducted separately to explore their perspectives on the process implementation of the SIMSP according to their roles and responsibilities. A topic guide with open-ended questions are developed and use in the FGD to get feedback on the appropriateness, feasibility (facilitators and barriers), effectiveness, and recommendations for improvement on the SIMSP.

Statistical Analysis:

Data analysis is conducted using SPSS version 24 software, and Qualitative Data Analysis Software (NVivo) version 11 software.

Descriptive Analysis:

The frequency distribution, a measure of central tendency and dispersion are carried out. Continuous data are presented in mean and standard deviation (or median and interquartile range) based on the normality of the data. Categorical data are presented in frequency and percentages. The demographics of the sample are analysed using descriptive statistics.

Effectiveness Analysis:

Intention to Treat (ITT) analysis will be applied to measure the effect of the SIMSP on the primary and secondary outcome measures over and above that by the usual care. Pearson Chi Square test is used to assess differences in the proportion of children with plaque between groups at baseline and after 6 months. Independent sample T-test is used to assess the difference in mean decrement plaque scores after 6 months between groups, and Paired sample T-test was used to assess within-group changes. Effect size of the SIMSP is calculated. Similar statistical tests are used to assess the differences in parental OHL between the groups after 6 months. For children's OHB, Pearson Chi Square test is used to assess differences in children's OHB between groups at baseline and after 6 months, while McNemar test is used for within-group changes in proportions.

ELIGIBILITY:
Inclusion Criteria:

* Children who are healthy
* Preschool children who can understand Malay language
* Parents who can speak and write in Malay language

Exclusion Criteria:

* Children with chronic medical conditions, dental/oral developmental conditions, long term medications, and physical disability

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 653 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-11-17 (Actual)

PRIMARY OUTCOMES:
The mean decrement in plaque score assessed using the Oral Cleanliness Index | 6 months
  The mean decrement in plaque score from baseline to follow up between the intervention and control group will be assessed. Assessment for the presence of visible plaque will involve examining the labial surfaces of upper right to upper left primary canines. Each of the surface is assessed by scoring; 0 = teeth appear clean, 1 = a little plaque visible (existence of plaque around the labial cervical margins and covering < ½ of labial tooth surfaces), 2 = substantial amount of plaque visible (plaque covering > ½ labial tooth surfaces), and 9 = assessment cannot be made (there is no teeth in both anterior segments for plaque assessment). Total score is the sum of scores from the 6 surfaces. Mean decrement score is obtained by subtracting mean score at follow up from mean score at baseline. Finally, mean decrement scores of intervention and control group are compared.

SECONDARY OUTCOMES:
Changes in child's oral health behaviours assessed using a self-reported questionnaire by parents | 6 months
  Changes in the prevalence of good oral health behaviours. The changes are recorded as follows: Brushing teeth with fluoride toothpaste (yes, no), tooth brushing frequency (at least 2x/day, < 2x/day), frequency of monitoring child's tooth brushing (daily, do not monitor), bottle feeding (yes, no), bottle feeding frequency (daily, infrequent), bottle feeding at night (yes, no), sugar intake (up to 4x/day, > 5x/day), dental visit (< 1 yr, between 1-2 yr, > 2 yr)
The mean increment of oral health literacy score of parents/guardians assessed using The Dental Health Literacy Assessment Index (DHLAI) | 6 months
  The DHLAI consists of 3 domains; (a) Oral Health Knowledge domain (12 items). Each item is assessed by one correct answer from 4 options. Total score = sum scores of correct answers with score range from 0-12; (b) Comprehension domain (5 items). Each item is scored by true/false answer options. Total score = the sum scores of correct answers with score range from 0-5; (c) Skills and Motivation domain (39 items). Each item is assessed using a 5-point Likert scale (strongly disagree to strongly agree). Total score = sum scores of all items with score range from 0-39. Total score of OHL = sum of scores from the 3 domains with score range from 0-56. Mean increment scores of total OHL and the 3 domains are calculated by subtracting the respective scores at baseline from follow up scores. The mean scores were compared between intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Zamros YM Yusof, BDS, MSc, PhD, Principal Investigator — Faculty of Dentistry, University of Malaya, Kuala Lumpur, 50603, Malaysia
Locations (1):
- State Education Department, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No
Data will be kept at the Faculty of Dentistry, University of Malaya, 50603, Kuala Lumpur, Malaysia. Data can be shared upon request and is subjected to the data protection regulations.

REFERENCES:
- [Background] Albino J, Tiwari T. Preventing Childhood Caries: A Review of Recent Behavioral Research. J Dent Res. 2016 Jan;95(1):35-42. doi: 10.1177/0022034515609034. Epub 2015 Oct 5. PMID 26438210
- [Background] Bearn DR, Aird JC, Jenkins WM, Kinane DF. Index of Oral Cleanliness (I.O.C.). A new oral hygiene index for use in clinical audit. Br J Orthod. 1996 May;23(2):145-51. doi: 10.1179/bjo.23.2.145. PMID 8771339
- [Background] Cooper AM, O'Malley LA, Elison SN, Armstrong R, Burnside G, Adair P, Dugdill L, Pine C. Primary school-based behavioural interventions for preventing caries. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD009378. doi: 10.1002/14651858.CD009378.pub2. PMID 23728691
- [Background] Freeman, R, Gibson, B, Humphris, GM, Leonard, H, Yuan, S & Whelton, H. School-based health education programmes, health-learning capacity and child oral health-related quality of life. Health Education Journal. 2016;75(6):698-711.
- [Background] Gao X, Lo EC, McGrath C, Ho SM. Innovative interventions to promote positive dental health behaviors and prevent dental caries in preschool children: study protocol for a randomized controlled trial. Trials. 2013 Apr 30;14:118. doi: 10.1186/1745-6215-14-118. PMID 23782918
- [Background] Guse K, Levine D, Martins S, Lira A, Gaarde J, Westmorland W, Gilliam M. Interventions using new digital media to improve adolescent sexual health: a systematic review. J Adolesc Health. 2012 Dec;51(6):535-43. doi: 10.1016/j.jadohealth.2012.03.014. Epub 2012 May 5. PMID 23174462
- [Background] Marinho VC, Higgins JP, Sheiham A, Logan S. Fluoride toothpastes for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2003;2003(1):CD002278. doi: 10.1002/14651858.CD002278. PMID 12535435
- [Background] Mejare I, Axelsson S, Dahlen G, Espelid I, Norlund A, Tranaeus S, Twetman S. Caries risk assessment. A systematic review. Acta Odontol Scand. 2014 Feb;72(2):81-91. doi: 10.3109/00016357.2013.822548. Epub 2013 Sep 2. PMID 23998481
- [Background] Peretz B, Ram D, Azo E, Efrat Y. Preschool caries as an indicator of future caries: a longitudinal study. Pediatr Dent. 2003 Mar-Apr;25(2):114-8. PMID 12723835
- [Background] Pine CM. Designing school programmes to be effective vehicles for changing oral hygiene behaviour. Int Dent J. 2007;57(S5):377-81.
- [Background] Rajab LD, Petersen PE, Bakaeen G, Hamdan MA. Oral health behaviour of schoolchildren and parents in Jordan. Int J Paediatr Dent. 2002 May;12(3):168-76. doi: 10.1046/j.1365-263x.2002.00359.x. PMID 12028308
- [Background] Sheiham A. Dietary effects on dental diseases. Public Health Nutr. 2001 Apr;4(2B):569-91. doi: 10.1079/phn2001142. PMID 11683551
- [Background] Songur F, Simsek Derelioglu S, Yilmaz S, Kosan Z. Assessing the Impact of Early Childhood Caries on the Development of First Permanent Molar Decays. Front Public Health. 2019 Jul 9;7:186. doi: 10.3389/fpubh.2019.00186. eCollection 2019. PMID 31338357
- [Background] Pitts NB, Ekstrand KR; ICDAS Foundation. International Caries Detection and Assessment System (ICDAS) and its International Caries Classification and Management System (ICCMS) - methods for staging of the caries process and enabling dentists to manage caries. Community Dent Oral Epidemiol. 2013 Feb;41(1):e41-52. doi: 10.1111/cdoe.12025. PMID 24916677
- [Background] . Ludke RL, Kudel I, and Weber DL, Dental Health Literacy Assessment Instrument, U.o. Cincinnati, Editor. 2008.
- [Derived] Yusof ZYM, Anwar NH, Mohd Nor NA, Nor MM, Mustafa SE. The effect of the SIMS Programme versus existing preschool oral healthcare programme on oral hygiene level of preschool children: study protocol for a cluster randomised controlled trial. Trials. 2021 Feb 22;22(1):156. doi: 10.1186/s13063-021-05111-0. PMID 33618735
- See also: National Oral Health Survey of Preschool Children, Malaysia, 2015 — http://irep.iium.edu.my/62539/